CLINICAL TRIAL: NCT00214981
Title: A 1-Year, Open-Label, Flexible-Dosage Study to Evaluate the Safety and Continued Efficacy of Modafinil (Film-coated Tablet Formulation) in Children and Adolescents With Attention-Deficit/Hyperactivity Disorder (Followed by an Open-Ended Extension Period)
Brief Title: Evaluate the Safety and Efficacy of Modafinil in Children and Adolescents With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1538D/312/AD/US
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Attention Deficit/Hyperactivity Disorder; ADHD
Keywords: ADHD; Attention Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Modafinil

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
Primary objective of this study is to evaluate the safety of treatment with modafinil film-coated tablet.

ELIGIBILITY:
Inclusion Criteria: Patients are included in the study if they participated in a previous qualifying study with modafinil and, in the opinion of the investigator, will continue to benefit from treatment with modafinil. In addition, the following criteria must be met:

* a boy or girl 6 to 17 years of age, inclusive, and English-speaking
* weight and height between the 5th and 95th percentile on the National Center for Health Statistics (NCHS) growth chart for age, height, and weight
* if more than 6 months since last dose of study drug, meets the full DSM-IV crieria for ADHD (combined typd, predominantly inattentive type, or predominantly hyperactive - impulsive type) at screening, as manifested by a psychiatric/clinical evaluation and confirmed by a structured diagnostic interview, namely, the Diagnostic Interview Schedule for Children, Fourth Edition (DISC-IV).
* are in good health (except for a diagnosis of ADHD) as determined by medical and psychiatric history, physical examination, ECG, serum chemistry, hematology, urinalysis
* girls of child bearing potential (Tanner scale >3) OR all girls 8 years of age and older have a negative urine pregnancy test at screening, must be using a medically acceptable method of birth control, and must agree to continue use of this method for the duration of the study (and for 30 days after participation in the study). (NOTE: For conducting pregnancy tests, the investigator has the option of determining the sexual maturity all girls 8 years of age and older.) Acceptable methods of birth control include: barrier method with spermicide; steroidal contraceptive (eg, oral, transdermal, implanted, and injected) in conjunction with a barrier method; intrauterine device (IUD); or abstinence
* have a parent or legal guardian who is willing to participate in the study.

Exclusion Criteria: Patients are excluded from participating in this study if 1 or more of the following criteria are met:

* a history or current diagnosis of pervasive developmental disorder, schizophrenia, or other psychotic disorders, or a clinical assessment of current suicide risk
* any current psychiatric comorbidity, including but not limited to depression or other mood disorder, anxiety disorder, or pervasive mental disorder, that requires pharmacotherapy
* a clinically significant drug sensitivity to stimulants such as amphetamine, dextroamphetamine, methylphenidate, pemoline
* failure to respond to 2 or more adequate courses (dose or duration) of ADHD therapy
* use of any other prescription medications for ADHD (e.g., amphetamine, dextroamphetamine, methylphenidate, pemoline, atomoxetine) after the screening visit
* use of any MAO inhibitors or SSRIs within 2 weeks of the baseline visit
* hypertension, defined as follows (SBP = systolic blood pressure and DBP = diastolic blood pressure):
* ages 6-9 years SBP > 122mmHg or DBP>78mmHg
* ages 10-12 years SBP > 126mmHg or DBP>82mmHg
* ages 13-17 years SBP > 136mmHg or DBP>86mmHg
* hypotension, defined as sitting systolic blood pressure (taken after resting for 5 minutes) of less than 50mmHg for children under 12 years of age or less than 80mmHg for children 12 and older
* a sitting pulse outside the range of 60 through 115 bpm after resting for 5 minutes

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2003-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of treatment with the modafinil film coated tablet.

CONTACTS AND LOCATIONS:
Locations (57):
- United States (57):
  - University of Alabama Birmingh, Birmingham, Alabama
  - Pivotal Research Center, Mesa, Arizona
  - River Valley Neurology, Fort Smith, Arkansas
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - UCI Child Development Center, Irvine, California
  - BMR HealthQuest, San Diego, California
  - University of CA San Francisco, San Francisco, California
  - Encompass Clinical Research, Spring Valley, California
  - Alpine Clinical Research, Boulder, Colorado
  - Sarkis Clinical Trials, Gainesville, Florida
  - Amedica Research Inst., Hialeah, Florida
  - Children's Developmental Cente, Maitland, Florida
  - Miami Research Associates, Miami, Florida
  - Clinical Neuroscience Solution, West Palm Beach, Florida
  - Child Neurology Assoc., Atlanta, Georgia
  - Mountainview Center for Resear, Decatur, Georgia
  - Foothills Psychiatry, Boise, Idaho
  - Consultants in Neurology, Ltd., Northbrook, Illinois
  - Midwest Neurology, Inc., Danville, Indiana
  - Cientifica at Prarie View, Newton, Kansas
  - Vince and Associates Clinical, Overland Park, Kansas
  - Kentucky Pediatric/Adult Resea, Bardstown, Kentucky
  - Michael J. Rieser, MD, Lexington, Kentucky
  - Pedia Research, LLC, Owensboro, Kentucky
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Dolby Providers, Inc., New Orleans, Louisiana
  - NeuroScience, Inc., Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Clinical Neurophysiology Svcs, Troy, Michigan
  - University of Nebraska, Omaha, Nebraska
  - Clinical Research Center of NV, Las Vegas, Nevada
  - Radiant Research Las Vegas, Las Vegas, Nevada
  - CNS Research Institute, Clementon, New Jersey
  - Children's Specialized Hospita, Toms River, New Jersey
  - University of Buffalo, Buffalo, New York
  - New York Psychiatric Inst, New York, New York
  - University of Rochester, Rochester, New York
  - North Carolina Neuropsychiatry, Chapel Hill, North Carolina
  - North Carolina Neuropsychiatry, Charlotte, North Carolina
  - Psychiatric Professional Servi, Cincinnati, Ohio
  - Pahl Pharmaceutical Research, Oklahoma City, Oklahoma
  - OCCI Eugene, Eugene, Oregon
  - Summit Research Network Inc., Portland, Oregon
  - OCCI, Inc., Salem, Oregon
  - CNS Research Institute PC, Philadelphia, Pennsylvania
  - Primary Physicians Research, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Clinical Neuroscience Solution, Memphis, Tennessee
  - Vanderbilt University Medical, Nashville, Tennessee
  - Dallas Pediatric Neurology, Dallas, Texas
  - UT Health Science Center, San Antonio, Texas
  - Radiant Research Salt Lake, Salt Lake City, Utah
  - Otter Creek Clinical Studies, Burlington, Vermont
  - Monarch Research Associates, Norfolk, Virginia
  - James A. Knutson, MD, Kirkland, Washington
  - Pacific Institute of Mental He, Seattle, Washington
  - Marshfield Clinical Research, Marshfield, Wisconsin